CLINICAL TRIAL: NCT05737082
Title: A Randomized, Open Label, Single Dose, 4-period Replicate Crossover Clinical Trial to Evaluate the Pharmacokinetic Characteristics and Safety After Administration of a Fixed-dose Combination Drug of HCP2201 and Co-administration of RLD2205 and RLD2206 in Healthy Male Volunteers Under Fasting Conditions
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety Between HCP2201 and Co-administration of Each Component in Healty Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-PRADA-101
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): * Period 1, Period 3: RLD2205 + RLD2206
  * Period 2, Period 4: HCP2201
  Interventions: Drug: HCP2201; Drug: RLD2205; Drug: RLD2206
- Sequence 2 (Experimental): * Period 1, Period 3: HCP2201
  * Period 2, Period 4: RLD2205 + RLD2206
  Interventions: Drug: HCP2201; Drug: RLD2205; Drug: RLD2206

INTERVENTIONS:
Drug: HCP2201 — Take 2 tablets once per period
Drug: RLD2205 — Take 2 tablets once per period
Drug: RLD2206 — Take 1 tablet once per period

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic characteristics and safety between HCP2201 and co-administration of each component in fasting condition in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 19~55 years in healthy male volunteers
* 19 kg/m^2 ≤ BMI < 28 kg/m^2, weight ≥55kg
* 90 mmHg ≤ SBP <140 mmHg, 50 mmHg ≤ DBP <90 mmHg
* Agrees that the person, spouse, or partner uses appropriate medically recognized contraception and does not provide sperm from the date of administration of the first investigational drug to 7 days after the administration of the last investigational drug.
* Subjects who voluntarily decides to participate in this clinical trial and agree in writing to ensure compliance with the clinical trial

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
* Subjects who judged ineligible by the investigator

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-05-14 (Actual)

PRIMARY OUTCOMES:
Abiraterone acetate AUCt | 0~72 hours
  Pharmacokinetic evaluation
Abiraterone acetate Cmax | 0~72 hours
  Pharmacokinetic evaluation
Prednisolone AUCt | 0~24 hours
  Pharmacokinetic evaluation
Prednisolone Cmax | 0~24 hours
  Pharmacokinetic evaluation

SECONDARY OUTCOMES:
AUCinf | 0~72 hours
  Pharmacokinetic evaluation
Tmax | 0~72 hours
  Pharmacokinetic evaluation
t1/2 | 0~72 hours
  Pharmacokinetic evaluation
CL/F | 0~72 hours
  Pharmacokinetic evaluation
Vd/F | 0~72 hours
  Pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Min-gul Kim, MD, Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea